CLINICAL TRIAL: NCT03899597
Title: A Prospective, Randomized and Placebo Controlled Trial Comparing the Role of ARTificial Uterine CONtractions and no Intervention in Perinatal Respiratory Morbidity of Term Infants Delivered by Elective Caesarean Section - ARTCON Study
Brief Title: The Role of ARTificial Uterine CONtractions in Perinatal Respiratory Morbidity of Term Infants Delivered by Elective Caesarean Section
Acronym: ARTCON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute for the Care of Mother and Child, Prague, Czech Republic (Other)
Responsible Party: Principal Investigator, Ivan Berka, Head of Neonatal Intensive Care Unit, Institute for the Care of Mother and Child, Prague, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ARTCON Study Protocol
Record Dates: First submitted 2019-03-31; First posted 2019-04-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Neonatal Respiratory Distress
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Oxytocin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- artificial contractions (ARTCON) group (Experimental): All participating patients in the intervention (ARTCON) group will undergo oxytocin exposure in the form of a continuous intravenous infusion according to dosage guidelines of The Czech Society of Obstetrics and Gynaecology. The exposure will take two hours to complete and should be finished at least one hour before elective caesarean section is performed in order for the assumed effects of physiological stress associated with labor to occur.
  Interventions: Drug: Oxytocin
- standard approach (SA) group (Placebo Comparator): All participating patients in the control (SA) group will undergo placebo exposure in the form of a continuous intravenous infusion. The exposure will take two hours to complete and should be finished at least one hour before elective caesarean section is performed.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Oxytocin — The intervention group (ARTCON) will receive the standard assignment for the elective caesarean section, but at least one hour before surgery oxytocin exposure will be performed with cardiotocographic (CTG) monitoring and obstetrical supervision.
  Arms: artificial contractions (ARTCON) group
Other: Normal saline — The control group (SA) will receive the standard assignment for the elective caesarean section, but at least one hour before surgery placebo exposure will be performed with cardiotocographic (CTG) monitoring and obstetrical supervision.
  Other Names: Placebo
  Arms: standard approach (SA) group

SUMMARY:
In this study, the investigators aim to investigate if artificial uterine contractions prior to elective caesarean section delivery may have an impact on the respiratory morbidity of term neonates.

DETAILED DESCRIPTION:
Accumulating evidence suggests that the respiratory morbidity of infants is lower if delivered by caesarean section after the spontaneous onset of uterine contractions, or after oxytocin exposure. Moreover, benefits for the mother due to stretching of the lower uterine segment and possible lower blood loss are plausible.

In obstetrics, there is a well described and standardized way to induce artificial uterine contractions in order to predict fetal wellbeing and tolerance of labor, without inducing the labor itself. This is the oxytocin challenge test (OCT). Although the OCT has not been performed previously in the context of planned elective caesarean section deliveries, it is generally considered a safe procedure if appropriate monitoring is granted. Hence evaluation of the role of artificial uterine contractions in perinatal respiratory morbidity of term infants delivered by elective caesarean section is possible and of interest.

ELIGIBILITY:
Inclusion Criteria:

* Term/near-term pregnancy (36+0 - 41+6 weeks of gestation)
* Planned delivery by elective caesarean section
* Absence of any exclusion criteria
* Informed consent obtained

Exclusion Criteria:

* Term premature rupture of membranes (TPROM)
* Spontaneous onset of uterine contractions
* Known serious congenital malformations
* Placenta praevia/vasa praevia
* Abnormal placental attachment
* Intrauterine growth restriction (birth weight below 3rd centile for given gestational age and gender)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of neonatal respiratory morbidity | First 24 hours after delivery
  Neonatal respiratory morbidity during the first 24 hours after delivery is defined as presence of transitory tachypnoea of the newborn, or respiratory distress syndrome, and/or persistent pulmonary hypertension of the newborn.

SECONDARY OUTCOMES:
Oxytocin challenge test effectivity | Before elective caesarean section
  Contractions being induced (felt or CTG recorded) before elective caesarean section
Oxytocin challenge test safety and feasibility | Before elective caesarean section
  CTG trace suggestive of hypoxia during oxytocin exposure. Subjectively unbearable pain and discomfort during oxytocin exposure.
Maternal blood loss | During caesarean section
  Defined as the difference in hemoglobin levels before and after surgery
Total duration of surgery | Time of caesarean section
  Minutes
Lamellar body count in amniotic fluid | During caesarean section
  Particles per microlitre
Incidence of transitory tachypnoea of the newborn | First 24 hours after delivery
  Breathing rate above 60 per minute at least for 3 hours (3 consecutive measurements) and /or dyspnoea for at least two hours in the follow-up period (consecutive) and /or the need for oxygen therapy during the first 24 hours after birth.
Incidence of respiratory distress syndrome | First 24 hours after delivery
  Defined by need for ventilatory support in the first 24 hours after birth (nasal continuous positive airway pressure, mechanical ventilation) and X-ray examination results consistent with RDS diagnosis.
Incidence of perinatal hypoxia | First 24 hours after delivery
  Presence of diagnostic criteria of hypoxic-ischaemic encephalopathy: 5-min Apgar score of less than 5, need for delivery room intubation or CPR, umbilical cord arterial pH less than 7.00 and abnormal neurological signs such as hypotonic muscles or lack of sucking reflex
Incidence of early onset sepsis | First 48 hours after delivery
  Clinical or proven (positive blood culture)
Incidence of significantly increased neonatal pulmonary vascular resistance | First 72 hours after delivery
  Pulmonary vascular resistance measurements consist of measuring the right ventricular systolic pressure (RVSP), pulmonary artery pressure (PAP) and persistent ductus arteriosus (PDA) shunting (if present).
Incidence of persistent pulmonary hypertension of the newborn | First 24 hours after delivery
  Defined by marked pulmonary hypertension that causes hypoxemia secondary to right-to-left shunting of blood at the foramen ovale and ductus arteriosus.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Berka, MD, Principal Investigator — Institute for the Care of Mother and Child, Prague, Czech Republic
Locations (1):
- Institute for the Care of Mother and Child, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No